CLINICAL TRIAL: NCT03305120
Title: Musculo-scrawny Manifestation Associated With the Endometriosis
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: ENDOMETRI-OS
Record Dates: First submitted 2017-10-04; First posted 2017-10-09 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: pain VAS evaluation — each patient has to answer to a questionnaire about pain

SUMMARY:
The endometriosis is defined by the presence of endometriosic tissue outside of the womb and the prevalence is estimated to be 10% of women.Here is a project aimed to compare musculo-scrawny pains between patients with endometriosis and whose don't suffer of this pathology;

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 45
* consulting in Service of gynecology
* First trimester of pregnancy or for pap smears

Exclusion Criteria:

* endometriosis diagnostic already done
* rhumalogic disease known
* age < 18 and > 50
* menopause

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — only women
Study Population: patient consulting in gynecologic service of GHPSJ
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2016-09-16 (Actual); Primary Completion 2016-10-16 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
VAS of musculo-scrawny pain | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France